CLINICAL TRIAL: NCT00734305
Title: A Phase I and Pharmocologic Study of MM-121 in Patients With Refractory Advanced Solid Tumors
Brief Title: Phase I Safety Study of the Drug MM-121 in Patients With Advanced Solid Tumors Resisting Ordinary Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-121-01-100; MM-121
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Solid Tumors
Keywords: cancer, solid tumors, oncology, Phase I, ErbB3, HER3; (erbB-3, HER-3)
MeSH Terms: conditions — Neoplasms; Lethal Congenital Contracture Syndrome 2 | interventions — seribantumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental): Cohorts of escalating doses of MM-121 administered IV QW to determine MTD or RP2D + expansion cohort at MTD/RP2D
  Interventions: Drug: MM-121

INTERVENTIONS:
Drug: MM-121 — Dose escalation Frequency - once weekly
  Other Names: Seribantumab, SAR256212

SUMMARY:
This study was a Phase 1 and pharmacologic open-labeled dose-escalation trial using a "3+3" design to determine maximum tolerated dose/recommended Phase 2 dose.

DETAILED DESCRIPTION:
Successive cohorts of three or more patients were treated at escalating doses until a maximum tolerated dose/recommended phase 2 dose was identified. The study initially explored a dosing schedule every 7-days, which may have been modified to longer intervals under certain circumstances but did not expand to more than weekly. When the maximum tolerated dose/recommended Phase 2 dose was identified, an Expansion Cohort was enrolled at that dose to further characterize safety and to explore pharmacodynamic endpoints. There were 3 sites that participated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced solid tumors that have recurred or progressed following standard therapy, or that have not responded to standard therapy, or for which there is no standard therapy, or who are not candidates for standard therapy
* Patients must be > 18 years of age
* Patients or their legal representatives must be able to understand and sign an informed consent form
* Patients must have evaluable or measurable tumor(s)

  * Patients must be recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy. Up to CTCAE Grade 1 is acceptable for patients with known peripheral neuropathy.
  * Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-121 (an effective form of contraception is an oral contraceptive or a double barrier method)

In addition, patients to be enrolled the Expansion Cohort must have/be:

* Advanced/metastatic breast cancer with histological/cytological documentation of ER-, PR-, Her2/neu non-over-expressing breast cancer (triple negative breast cancer); OR,
* Patients must have advanced/metastatic breast cancer with histologically or cytologically confirmed ER+ and/or PR+, Her2/neu non-over-expxressing OR,
* Patients must have advanced/metastatic histological confirmation of epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer; OR,
* Additional tumor types such as metastatic colorectal, advanced non small cell lung cancer, and others may be considered on a per-patient basis
* Tumor tissue amenable to biopsy
* Platelet counts, partial thromboplastin time (PTT) and international normalized ratio (INR) within normal limits.
* Willing to undergo tumor biopsy twice (once before and once after treatment with MM-121)
* Blocks of archived formalin-fixed, paraffin-embedded, unstained tumor tissue available for submission. Patients with no available archived tumor tissue available must receive Sponsor approval prior to enrollment.

Exclusion Criteria:

* Patients for whom potentially curative antineoplastic therapy is available
* Patients who are pregnant or lactating
* Patients with an active infection or with an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing. (At the discretion of the investigator, patients with tumor fever may be enrolled.)
* Patients with untreated and/or symptomatic CNS malignancies (primary or metastatic); patients with CNS metastases who have undergone surgery or radiotherapy, whose disease is stable, and who have been on a stable dose of corticosteroids for at least 2 weeks prior to the first scheduled day of dosing will be eligible for the trial
* NYHA Class III or IV congestive heart failure or LVEF < 55%
* Known HIV, hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Denlinger, MD, Principal Investigator — Fox Chase Cancer Center; Kwok Kin Wong, MD, Principal Investigator — Dana-Farber Cancer Institute; Keedy L Vicki, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denlinger CS, Keedy VL, Moyo V, MacBeath G, Shapiro GI. Phase 1 dose escalation study of seribantumab (MM-121), an anti-HER3 monoclonal antibody, in patients with advanced solid tumors. Invest New Drugs. 2021 Dec;39(6):1604-1612. doi: 10.1007/s10637-021-01145-y. Epub 2021 Jul 11. PMID 34250553

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation: Cohort 1: MM-121: 3.2 mg/kg IV QW
- Dose Escalation: Cohort 2: MM-121: 6 mg/kg IV QW
- Dose Escalation: Cohort 3: MM-121: 10 mg/kg IV QW
- Dose Escalation: Cohort 4: MM-121: 15 mg/kg IV QW
- Dose Escalation: Cohort 5: MM-121: 20 mg/kg IV QW
- Dose Escalation: Cohort 6: MM-121: 40 mg/kg IV loading dose on C1W1 followed by weekly maintenance doses of 20 mg/kg IV QW
- Expansion Cohort: (Highest tested dose in absence of reaching maximum tolerated dose) 40 mg/kg IV loading dose on C1W1 followed by weekly maintenance doses of 20 mg/kg IV QW
Period: Overall Study
Arm/Group | Dose Escalation: Cohort 1 | Dose Escalation: Cohort 2 | Dose Escalation: Cohort 3 | Dose Escalation: Cohort 4 | Dose Escalation: Cohort 5 | Dose Escalation: Cohort 6 | Expansion Cohort
Started | 7 | 3 | 4 | 3 | 5 | 4 | 18
Completed | 6 (1 patient was enrolled but did not meet eligibility criteria at C1W1, and thus was never dosed) | 3 | 4 | 3 | 5 | 4 | 18
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MM-121 Dose Escalation: MM-121: Dose escalation Frequency - once weekly IV
- MM-121 Expansion Cohort: Expansion cohort at recommended phase 2 dose
- Total: Total of all reporting groups
Arm/Group | MM-121 Dose Escalation | MM-121 Expansion Cohort | Total
Number analyzed (Participants) | 25 | 18 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.82) | 58.5 (8.08) | 59.85 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 13 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 17 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 17 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate and Duration
Description: To determine the number of patients reporting an objective response using RECIST v 1.1 where a Partial Response is defined as a >20% decrease in tumor burden from baseline and a Complete Response is defined as complete disappearance of tumor burden from baseline. Duration of response is defined as the length of time in weeks from observation of response until progression.
  NOTE: because no patients experienced an objective response as shown below, duration of response is not presented. No duration of response could be measured.
Time Frame: Time from first dose to date of progression, with a median of 7.1 weeks
Measure: Number; unit: participants with objective response
Groups:
- Dose Escalation: Cohort 2: MM-121 6 mg/kg IV QW
- Dose Escalation: Cohort 3: MM-121 10 mg/kg IV QW
- Dose Escalation: Cohort 4: MM-121 15 mg/kg IV QW
- Dose Escalation: Cohort 5: MM-121 20 mg/kg IV QW
- Dose Escalation: Cohort 6: MM-121 40 mg/kg IV loading dose on Cycle 1, Week 1 followed by 20 mg/kg IV weekly maintenance doses
Arm/Group | Dose Escalation: Cohort 1 | Dose Escalation: Cohort 2 | Dose Escalation: Cohort 3 | Dose Escalation: Cohort 4 | Dose Escalation: Cohort 5 | Dose Escalation: Cohort 6 | MM-121 Expansion Cohort
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 5 | 4 | 18
participants with objective response | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Determine the Maximum Tolerated Dose Dependent on Reports of Dose-limiting Toxicities
Description: Using a 3+3 dose escalation model, the maximum tolerated dose was determined by assessing dose-limiting toxicities in each cohort from cohort 1-6. Cohort 1 began at 3.2 mg/kg IV QW and the dose escalated in separate cohorts from 6 mg/kg IV QW, 10 mg/kg IV QW, 15 mg/kg IV QW, 20 mg/kg IV QW, to the highest scheduled testing dose at 40 mg/kg one-time loading dose on cycle 1, week 1 followed by 20 mg/kg IV QW maintenance doses. If 3 patients were treated and passed the observation window, escalation to the next cohort was initiated. If a DLT was reported, 3-4 additional patients were enrolled and observed. If a DLT was observed in the expanded cohort, this dose was considered to be the maximum tolerated dose. The maximum tolerated dose was defined at the cohort in which two dose-limiting toxicities were observed, or as the highest target dose tested in the absence of DLTs. The determined MTD was considered the Recommended Phase 2 Dose and was used to open the expansion cohort.
Time Frame: From date of first dose to 30 days after termination, the longest 47 weeks
Population: All participants in the 6 cohorts of dose escalation
Measure: Number; unit: mg/kg
Groups:
- Dose Escalation: All Participants: MM-121: Dose escalation Frequency - once weekly
Arm/Group | Dose Escalation: All Participants
Number analyzed (Participants) | 25
mg/kg | 40

3. Secondary Outcome: To Describe the Dose-limiting Toxicity of MM-121 as a Monotherapy
Description: To establish the safety of escalating doses of MM-121 administered as a monotherapy in order to determine the recommended phase 2 dose. Dose-escalation conducted using standard 3+3 model to determine maximum tolerated dose. Reports of Dose-Limiting Toxicities (DLTs) were assessed to determine the MTD to be used for the expansion cohort. DLTs were not measured in the Expansion Cohort.
Time Frame: From date of first dose to 30 days after termination, the longest 47 weeks
Measure: Number; unit: participants reporting DLTs
Groups:
- Cohort 1: MM-121 3.2 mg/kg IV QW
- Cohort 2: MM-121: 6 mg/kg IV QW
- Cohort 3: MM-121: 10 mg/kg IV QW
- Cohort 4: MM-121: 15 mg/kg IV QW
- Cohort 5: MM-121: 20 mg/kg IV QW
- Cohort 6: MM-121: 40 mg/kg IV loading dose followed by 20 mg/kg IV QW maintenance doses
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 5 | 4
participants reporting DLTs | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: To Determine the Pharmacokinetic and Immunogenicity Parameters of MM-121
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. The maximum observed concentration (Cmax) is presented and was calculated usig Non-compartmental analysis (NCA). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (3.2 mg/kg, 6 mg/kg, 10 mg/kg, 15 mg/kg, 20 mg/kg, 40/20 mg/kg).
  Immunogenicity data is not available.
Time Frame: At Cycle 1, Week 1 pre-treatment, at the end of the infusion, and 2, 4, 8, 24, 48 and 72 hours after starting the infusion; pre-dose collections on Cycle 1, Week 2 and Cycle 2, Week 1 for all patients
Population: All patients. NOTE: There are 22 patients included in the final cohort (4 patients in dose escalation portion Cohort 6 + 18 patients in Expansion Cohort), as PK analysis was performed per dose level and not per cohort. Cohort 6 and the Expansion Cohort were administered the same dose, and therefore the analysis reflects all 22 patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- Recommended Phase 2 Dose: MM-121: 40 mg/kg IV loading dose followed by 20 mg/kg IV QW maintenance doses Combination of Cohort 6 patients (N=4) and Expansion Cohort Patients (N=18) that received this dose level.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Recommended Phase 2 Dose
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 5 | 22
ug/mL | 78.1 (16.7) | 291 (42.4) | 410 (40.7) | 409 (17.0) | 518 (26.2) | 836 (23.9)

5. Secondary Outcome: To Determine the Pharmacokinetic Parameters of MM-121
Description: Pharmacokinetic (PK) evaluation was performed on plasma samples obtained weekly for the first cycle of the study and then on day 1 of each additional cycle to assess pre-treatment trough concentrations of MM-121. The AUC is presented and was calculated usig Non-compartmental analysis (NCA). Serum levels of MM-121 were measured at a central lab using an enzyme-linked immunosorbent assay (ELISA). Data is presented per dose level of MM-121 (3.2 mg/kg, 6 mg/kg, 10 mg/kg, 15 mg/kg, 20 mg/kg, 40/20 mg/kg).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr* ug/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Recommended Phase 2 Dose
Number analyzed (Participants) | 6 | 3 | 4 | 3 | 5 | 22
hr* ug/mL | 4850 (24.5) | 14800 (43.8) | 24000 (40.4) | 28100 (19.9) | 32700 (23.6) | 65600 (22.9)

ADVERSE EVENTS:
Time Frame: AEs were collected from a patient's first dose until 30 days after treatment termination. SAEs were collected from time of informed consent until 30 days after termination. If related, events could be reported at any time after termination.
Description: All related AEs ongoing at the time of treatment discontinuation were followed until resolution. Investigators were to report any AEs/SAEs assumed to be related any time, even if occurring more than 30 days after last dose. Though different for each patient, on average, patients could be followed for related AEs/SAEs for ~1 year after termination.
Groups:
- All Participatants: Dose Escalation cohort participants + Expansion cohort participants
Arm/Group | All Participatants
Serious Adverse Events (participants affected / at risk) | 14/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participatants (N=43)
Disease Progression (General disorders) | 4
Pyrexia (General disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Ureteric Obstruction (Renal and urinary disorders) | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participatants (N=43)
Nausea (Gastrointestinal disorders) | 20 — Any Relationship
Diarrhea (Gastrointestinal disorders) | 16 — Any Relationship
Vomiting (Gastrointestinal disorders) | 12 — Any Relationship
Abdominal Pain (Gastrointestinal disorders) | 7 — Any Relationship
Dyspepsia (Gastrointestinal disorders) | 5 — Any Relationship
Constipation (Gastrointestinal disorders) | 4 — Any Relationship
Stomatitis (Gastrointestinal disorders) | 4 — Any Relationship
Decreased Appetite (Metabolism and nutrition disorders) | 12 — Any Relationship
Hypokalemia (Metabolism and nutrition disorders) | 11 — Any Relationship
Hyperglycemia (Metabolism and nutrition disorders) | 10 — Any Relationship
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 — Any Relationship
Dehydration (Metabolism and nutrition disorders) | 7 — Any Relationship
Hypomagnesemia (Metabolism and nutrition disorders) | 7 — Any Relationship
Hypocalcemia (Metabolism and nutrition disorders) | 6 — Any Relationship
Hyponatremia (Metabolism and nutrition disorders) | 4 — Any Relationship
Hemoglobin Decreased (Investigations) | 10 — Any Relationship
Weight Decreased (Investigations) | 9 — Any Relationship
Blood Alkaline Phosphatase Increased (Investigations) | 5 — Any Relationship
Aspartate Aminotransferase Increased (Investigations) | 4 — Any Relationship
Activated Partial Thrombostatin Time Prolonged (Investigations) | 3 — Any Relationship
Blood Creatinine Increased (Investigations) | 3 — Any Relationship
Ejection Fraction Decreased (Investigations) | 3 — Any Relationship
Electrocardiogram Qt Prolonged (Investigations) | 3 — Any Relationship
Fatigue (General disorders) | 21 — Any Relationship
Disease Progression (General disorders) | 4 — Any Relationship
Peripheral Edema (General disorders) | 4 — Any Relationship
Asthenia (General disorders) | 3 — Any Relationship
Chills (General disorders) | 3 — Any Relationship
Back Pain (Musculoskeletal and connective tissue disorders) | 6 — Any Relationship
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 — Any Relationship
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 — Any Relationship
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 — Any Relationship
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 — Any Relationship
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 — Any Relationship
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 — Any Relationship
Cough (Respiratory, thoracic and mediastinal disorders) | 3 — Any Relationship
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 — Any Relationship
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 — Any Relationship
Rash (Skin and subcutaneous tissue disorders) | 10 — Any Relationship
Dizziness (Nervous system disorders) | 4 — Any Relationship
Headache (Nervous system disorders) | 4 — Any Relationship
Anemia (Blood and lymphatic system disorders) | 5 — Any Relationship
Urinary Tract Infection (Infections and infestations) | 4 — Any Relationship
Hypotension (Vascular disorders) | 3 — Any Relationship

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less